CLINICAL TRIAL: NCT04918680
Title: Prospective Post-market Study Examining the Effectiveness of the EcoFit® Total Hip System With Implacross® E Polyethylene
Brief Title: Prospective Post-market Study Examining the Effectiveness of the EcoFit®
Status: Not yet recruiting | Type: Observational
Sponsor: Implantcast North America, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EcoFit® Post-market Study
Record Dates: First submitted 2021-05-13; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Degenerative Joint Disease; Femoral Fracture; Osteoarthritis, Hip; Traumatic Arthritis
MeSH Terms: conditions — Joint Diseases; Femoral Fractures; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- EcoFit® Total Hip System with implacross® E Polyethylene: Subjects who meet the indications for use for the EcoFit® Total Hip System with implacross® E Polyethylene and are candidates for a primary hip replacement.
  Interventions: Device: EcoFit® Total Hip System with implacross® E Polyethylene

INTERVENTIONS:
Device: EcoFit® Total Hip System with implacross® E Polyethylene — The EcoFit® Total Hip System is a primary hip replacement system indicated for patients who are candidates for a primary cementless hip replacement. implacross® E Polyethylene is one of the components in the EcoFit® system.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the EcoFit Hip with implacross E polyethylene for total hip replacement surgery.

DETAILED DESCRIPTION:
This study will assess the performance and success rate of the EcoFit Total Hip System. Survivorship and clinical outcomes will help determine implant success 36 months as defined by specific scoring systems and compared to other published data.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for a total primary hip replacement.
* Subject must have degenerative joint disease, including osteoarthritis or traumatic arthritis, OR a femoral fracture which can be treated by a primary hip replacement and no other hardware
* Subject has a BMI of 40.00 kg/m2 or less at the time of enrollment
* Subject is likely to be available for evaluation for the duration of the study
* Subject is able and willing to sign the informed consent and follow study procedures
* Subject is not pregnant

Exclusion Criteria:

* Subject has had a prior hip replacement in the subject hip
* Subject has an active cancer or is a survivor for <5 years except for squamous cell or basal cell skin cancer
* Subject has a chronic disease(s) where, in the opinion of the investigator, the disease will interfere with the patient's ability to follow the protocol
* Subject is currently a documented substance abuser (alcohol or other addictions)
* Subject has an infection, or history of infection (within the last 3 months), acute or chronic, local or systemic
* Subject has a history of muscular, neurological or vascular deficiencies which compromise the affected extremity
* Subject has a BMI > 40.00 kg/m2
* Subject has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is a prisoner
* Subject is pregnant
* Subject has known materials sensitivity (to metals)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PIs will recruit from their patient population; patients already intending to undergo a total hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-21 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Survival of the EcoFit Hip with implacross E polyethylene for total hip replacement surgery | 36 months
  Evaluate the overall survivorship of the devices. Observed product-related complications and revisions are recorded and documented.

SECONDARY OUTCOMES:
Evaluate the pre to post-op change in the Harris Hip Score | Pre-op, 6 months, 12 months, 24 months, 36 months
  The Harris Hip Score tracks pain, function/gait, performance in functional activities, and range of motion as interpreted by the surgeon. The responses determine a score which can be compared in different intervals.
Evaluate the pre to post-op change in the WOMAC Score | Pre-op, 6 months, 12 months, 24 months, 36 months
  The Western Ontario McMaster Arthritis Index, a questionnaire completed by the patient, tracks pain, stiffness, and difficulty with daily activities.
Device related complications | Through completion of study, an average of 3.5 years
  Detect any device related complications via the adverse events reporting

IPD SHARING:
Plan to Share IPD: Undecided